CLINICAL TRIAL: NCT01340443
Title: A Multi Centre, Single Arm, Observational Study on Safety and Efficacy of MabThera Plus Chemotherapy as 1st Line Treatment in Patients With DLBCL or FL
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) Plus Chemotherapy As First-Line Treatment in Patients With Diffuse Large B-Cell Lymphoma or Follicular Lymphoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25435
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the safety and efficacy of MabThera/Rituxan (rituximab) plus chemotherapy as first-line treatment in patients with diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL). Data will be collected from each patient during the 6 months of induction treatment and for up to 3 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20+ diffuse large B-cell lymphoma or follicular lymphoma
* Treatment with MabThera/Rituxan as per locally approved China package insert
* Documented patient with medical records

Exclusion Criteria:

* Previous treatment for diffuse large B-cell lymphoma or follicular lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated diffuse large B-cell lymphoma or follicular lymphoma patients
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2011-01-19 (Actual); Primary Completion 2016-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 4.5 years

SECONDARY OUTCOMES:
Overall Response Rate (complete response + partial response) | 4.5 years
Progression-free survival, defined as time from first treatment to lymphoma progression or death | 4.5 years
Overall Survival, defined as time from 1st treatment to death of any cause | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- China (24):
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - the First Hospital of Jilin University, Changchun
  - Xiangya Hospital of Centre-South University, Changsha
  - Changzhou First People's Hospital, Changzhou
  - Daqing Oilfield General Hospital, Daqing
  - The First People's Hospital of Foshan, Foshan
  - Fuzhou General Hospital, PLA Nanjing Military Area Command, Fuzhou
  - Fujian Provincial Hospital, Fuzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - The affiliated Hospital of Guiyang Medical College, Guiyang
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - Anhui Province Cancer Hospital, Hefei
  - Affiliated Hospital of Inner Mongolia Medical College, Hohhot
  - Shandong Cancer Hospital, Jinan
  - The First Affilliated Hospital of Kunming Medical College, Kunming
  - Lanzhou General Hospital, PLA Lanzhou Military Area Command, Lanzhou
  - Jiangsu Cancer Hospital, Nanjing
  - Hebei Medical University Fourth Hospital;(Tumor Hospital of Hebei Province), Shijiazhuang
  - Shanxi Province Cancer Hospital, Taiyuan
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - The Second Affiliated Hospital of The Fourth Military Medical University (Tangdu Hospital), Xi'an
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhongshan General Hospital, Zhongshan

REFERENCES:
- [Derived] Wu JQ, Song YP, Su LP, Zhang MZ, Li W, Hu Y, Zhang XH, Gao YH, Niu ZX, Feng R, Wang W, Peng JW, Li XL, Ouyang XN, Wu CP, Zhang WJ, Zeng Y, Xiao Z, Liang YM, Zhuang YZ, Wang JS, Sun ZM, Bai H, Cui TJ, Feng JF. Three-year Follow-up on the Safety and Effectiveness of Rituximab Plus Chemotherapy as First-Line Treatment of Diffuse Large B-Cell Lymphoma and Follicular Lymphoma in Real-World Clinical Settings in China: A Prospective, Multicenter, Noninterventional Study. Chin Med J (Engl). 2018 Aug 5;131(15):1767-1775. doi: 10.4103/0366-6999.237401. PMID 30058572
- [Derived] Wu J, Song Y, Su L, Xu L, Chen T, Zhao Z, Zhang M, Li W, Hu Y, Zhang X, Gao Y, Niu Z, Feng R, Wang W, Peng J, Li X, Ouyang X, Wu C, Zhang W, Zeng Y, Xiao Z, Liang Y, Zhuang Y, Wang J, Sun Z, Bai H, Cui T, Feng J. Rituximab plus chemotherapy as first-line treatment in Chinese patients with diffuse large B-cell lymphoma in routine practice: a prospective, multicentre, non-interventional study. BMC Cancer. 2016 Jul 26;16:537. doi: 10.1186/s12885-016-2523-7. PMID 27460571